CLINICAL TRIAL: NCT02708420
Title: Comparison of Hemodynamic Responses to Endotracheal Intubation With Glidescope Video Laryngoscope and Macintosh Direct Laryngoscope in Patients Undergoing Coronary Artery Bypass Surgery
Brief Title: Does Glidescope Video Laryngoscope is Related to Less Hemodynamic Response?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gata Haydarpasa Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GataHRH
Record Dates: First submitted 2016-02-27; First posted 2016-03-15 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2016-03

CONDITIONS: Blood Pressure
Keywords: Glidescope; Cardiovascular surgery; Macintosh Laryngoscope; Hemodynamic response; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glidescope intubation (Other): This standard GlideScope (GS) technique involves a midline laryngoscopy followed by insertion of a styletted endotracheal tube, once an adequate view of the vocal cords is achieved.
  Interventions: Device: Glidescope
- Macintosh Laryngoscope (Other): This standard technique involves laryngoscopy followed by insertion of a styletted endotracheal tube, once an adequate view of the vocal cords is achieved.
  Interventions: Device: Macintosh Laryngoscope

INTERVENTIONS:
Device: Glidescope — This standard GlideScope (GS) technique involves a midline laryngoscopy followed by insertion of a styletted endotracheal tube, once an adequate view of the vocal cords is achieved.
  Arms: Glidescope intubation
Device: Macintosh Laryngoscope — This technique involves a laryngoscopy followed by insertion of a styletted endotracheal tube, once an adequate view of the vocal cords is achieved.
  Arms: Macintosh Laryngoscope

SUMMARY:
Laryngoscopy and endotracheal intubation causes significant hemodynamic response and thus presents an increased risk for patients undergoing cardiac bypass surgery. Prevention or reduction of this increment is important for hemodynamic control. In this randomized single blind study, the aim of this study is to compare the hemodynamic responses of two different laryngoscopy techniques with Glidescope and Macintosh laryngoscope in coronary cardiac bypass surgery patients.

DETAILED DESCRIPTION:
Laryngoscopy and endotracheal intubation causes significant hemodynamic response and thus presents an increased risk for patients undergoing cardiac bypass surgery. Prevention or reduction of this increment is important for hemodynamic control. In this randomized single blind study, the aim of this study is to compare the hemodynamic responses of two different laryngoscopy techniques with Glidescope and Macintosh laryngoscope in coronary cardiac bypass surgery patients. After induction with our institutional protocol for cardiac bypass surgery, hemodynamic data including heart rate, systolic and diastolic arterial pressure data will be recorded. Time for intubation, age, sex, ASA status data will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical Status 2-3
* Patients undergoing elective cardiac bypass surgery

Exclusion Criteria:

* Difficult intubation history
* Need for Rapid sequence intubation or alternative intubation method
* Emergency procedures
* Patients that have predictive factors for difficult intubation
* Patients with permanent pacemaker

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-01-01; Primary Completion 2017-05-18 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 5 minutes; At start of laryngoscopy and after 30th seconds, 60th seconds, 90th seconds, 120th seconds, 3rd minutes, 4th minutes, 5th minutes
  invasive blood pressure (mmHg) monitoring
Change in heart rate | 5 minutes; At start of laryngoscopy and after 30th seconds, 60th seconds, 90th seconds, 120th seconds, 3rd minutes, 4th minutes, 5th minutes
  Heart rate (beats per minute) will be measured before induction, and throughout and after laryngoscopy
Change in diastolic blood pressure | 5 minutes; At start of laryngoscopy and after 30th seconds, 60th seconds, 90th seconds, 120th seconds, 3rd minutes, 4th minutes, 5th minutes
  invasive blood pressure (mmHg) monitoring
Change in mean arterial pressure | 5 minutes;At start of laryngoscopy and after 30th seconds, 60th seconds, 90th seconds, 120th seconds, 3rd minutes, 4th minutes, 5th minutes
  invasive blood pressure (mmHg) monitoring

SECONDARY OUTCOMES:
Procedure time | 10 minutes
  Total laryngoscopy and intubation time (minutes)
Cormack lehane laryngoscopic view will be recorded | 10 minutes
  laryngoscopic view data will be recorded according to Cormack Lehane scale (A Scale with 1-4)

CONTACTS AND LOCATIONS:
Overall Officials: Sezai Ozkan, Prof., Study Chair — Gata Haydarpasa Research Hospital
Locations (1):
- GATA Haydarpasa Training Hospital, Istanbul, Asia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Friedman Z, Gurevich L, Siddiqui N. The effect of a modified GlideScope intubation technique on procedure times, airway morbidity and haemodynamic response. Eur J Anaesthesiol. 2016 Mar;33(3):229-30. doi: 10.1097/EJA.0000000000000339. No abstract available. PMID 26760401
- [Background] Amini S, Shakib M. Hemodynamic changes following endotracheal intubation in patients undergoing cesarean section with general anesthesia: application of glidescope(R) videolaryngoscope versus direct laryngoscope. Anesth Pain Med. 2015 Mar 30;5(2):e21836. doi: 10.5812/aapm.21836. eCollection 2015 Apr. PMID 25866708
- [Background] Dashti M, Amini S, Azarfarin R, Totonchi Z, Hatami M. Hemodynamic changes following endotracheal intubation with glidescope((R)) video-laryngoscope in patients with untreated hypertension. Res Cardiovasc Med. 2014 May;3(2):e17598. doi: 10.5812/cardiovascmed.17598. Epub 2014 Apr 1. PMID 25478537
- [Background] Aqil M. A study of stress response to endotracheal intubation comparing glidescope and flexible fiberoptic bronchoscope. Pak J Med Sci. 2014 Sep;30(5):1001-6. doi: 10.12669/pjms.305.4788. PMID 25225515
- [Background] Pournajafian AR, Ghodraty MR, Faiz SH, Rahimzadeh P, Goodarzynejad H, Dogmehchi E. Comparing GlideScope Video Laryngoscope and Macintosh Laryngoscope Regarding Hemodynamic Responses During Orotracheal Intubation: A Randomized Controlled Trial. Iran Red Crescent Med J. 2014 Apr;16(4):e12334. doi: 10.5812/ircmj.12334. Epub 2014 Apr 5. PMID 24910788
- [Background] Maassen RL, Pieters BM, Maathuis B, Serroyen J, Marcus MA, Wouters P, van Zundert AA. Endotracheal intubation using videolaryngoscopy causes less cardiovascular response compared to classic direct laryngoscopy, in cardiac patients according a standard hospital protocol. Acta Anaesthesiol Belg. 2012;63(4):181-6. PMID 23610856
- [Background] Siddiqui N, Katznelson R, Friedman Z. Heart rate/blood pressure response and airway morbidity following tracheal intubation with direct laryngoscopy, GlideScope and Trachlight: a randomized control trial. Eur J Anaesthesiol. 2009 Sep;26(9):740-5. doi: 10.1097/EJA.0b013e32832b138d. PMID 19417675
- [Background] Xue FS, Zhang GH, Li XY, Sun HT, Li P, Li CW, Liu KP. Comparison of hemodynamic responses to orotracheal intubation with the GlideScope videolaryngoscope and the Macintosh direct laryngoscope. J Clin Anesth. 2007 Jun;19(4):245-50. doi: 10.1016/j.jclinane.2006.11.004. PMID 17572317
- [Background] Russell T, Khan S, Elman J, Katznelson R, Cooper RM. Measurement of forces applied during Macintosh direct laryngoscopy compared with GlideScope(R) videolaryngoscopy. Anaesthesia. 2012 Jun;67(6):626-31. doi: 10.1111/j.1365-2044.2012.07087.x. Epub 2012 Feb 21. PMID 22352799